CLINICAL TRIAL: NCT02369653
Title: A Phase III Randomized, Open Label, Multi-center Study of the Safety and Efficacy of Apixaban for Thromboembolism Prevention Versus No Systemic Anticoagulant Prophylaxis During Induction Chemotherapy in Children With Newly Diagnosed Acute Lymphoblastic Leukemia (ALL) or Lymphoma (T or B Cell) Treated With Asparaginase
Brief Title: A Study of the Safety and Effectiveness of Apixaban in Preventing Blood Clots in Children With Leukemia Who Have a Central Venous Catheter and Are Treated With Asparaginase
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CV185-155; 2014-000328-47 (EudraCT Number)
Record Dates: First submitted 2015-01-21; First posted 2015-02-24 (Estimated); Results first posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Lymphoma; Acute Lymphoblastic Leukemia
Keywords: Anticoagulation
MeSH Terms: conditions — Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Apixaban (Experimental): Children aged 1 to <18 years weighing 6 to <35 kg randomized to apixaban will receive a fixed dose apixaban based on body weight tier twice a day for approximately 28 days.
  Children aged 1 to <18 years weighing ≥ 35 kg will receive 2.5 mg of apixaban twice a day for approximately 28 days. Subjects ≥ 5 years may be administered either 2.5-mg, 0.5-mg tablets or oral solution apixaban. Subjects < 5years and < 35 kg may be administered 0.5-mg tablets only
  Interventions: Drug: Apixaban
- No systemic anticoagulant prophylaxis (Placebo Comparator): No systemic anticoagulant prophylaxis
  Interventions: Other: No systemic anticoagulant prophylaxis

INTERVENTIONS:
Drug: Apixaban
  Arms: Apixaban
Other: No systemic anticoagulant prophylaxis
  Arms: No systemic anticoagulant prophylaxis

SUMMARY:
The purpose of this study is to compare the effect of a blood thinning drug called Apixaban versus no administration of a blood thinning drug, in preventing blood clots in children with leukemia or lymphoma. Patients must be receiving chemotherapy, including asparaginase, and have a central line (a catheter inserted for administration of medications and blood sampling)

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* New diagnosis of de novo ALL, lymphomas (T or B cell), or mixed-phenotype acute leukemia
* Planned 3-4 drug systemic induction chemotherapy with a corticosteroid, vincristine and a single dose or multiple doses of asparaginase, with or without daunorubicin
* Functioning Central Venous Access Device
* Must be able to tolerate oral medication or have it administered via an Nasogastric tube (NGT) or GT tube
* Males and females,age 1 year(365 days) to < 18 (17 years and 364 days) years.

Exclusion Criteria:

* Subjects scheduled to have > 3 Lumbar Punctures over the course of the study treatment period
* Prior history of documented DVT or PE in the past 3 months
* Known inherited bleeding disorder or coagulopathy
* Major surgery [excluding Central Venous Access Device (CVAD) replacement and bone marrow aspiration and non-open biopsy] within the last 7 days prior to enrollment that may be associated with a risk of bleeding. Open biopsy is considered a major surgery.
* Uncontrolled severe hypertension at enrollment. Severe hypertension is defined as a systolic or diastolic blood pressure (BP) > 5 mm Hg above the 95th percentile as defined by the National High Blood Pressure Education Program Working Group (NHBPEP) established guidelines for the definition of normal and elevated blood pressure in children
* Extreme hyperleukocytosis, white blood cell (WBC) counts over 200 x 109/L (200,000/microL) at the time of enrollment
* Liver dysfunction manifested by SGTP (ALT) > 5X Upper limit of normal (ULN) and/or Aspartate aminotransferase (AST) >5 X ULN and/or direct (conjugated) bilirubin > 2X ULN
* Renal function < 30% of normal for age and size as determined by the Schwartz formula
* International normalized ratio (INR) > 1.4 and activated partial thromboplastin time (aPTT) > 3 seconds above the upper limit of normal for age, within 1 week prior to enrollment.
* History of allergy to apixaban or Factor Xa inhibitors
* History of significant adverse reaction or major bleeding related adverse reaction to other anticoagulant or antiplatelet agents
* History of any significant drug allergy (such as anaphylaxis or hepatotoxicity
* Any investigational drug being administered during the study

Other protocol inclusion/exclusion criteria may apply

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 512 (Actual)
Dates: Start 2015-10-22 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (92):
- United States (64):
  - Phoenix Children'S Hospital/Ctr. For Cancer & Blood Ctr., Phoenix, Arizona
  - City of Hope, Duarte, California
  - Loma Linda University Cancer Center, Loma Linda, California
  - Childrens Hospital Of La, Los Angeles, California
  - Children'S Hospital Of Orange County, Orange, California
  - Lucile Packard Children's Hospital (LPCH), Palo Alto, California
  - Rady Children'S Hospital - San Diego, San Diego, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University School Of Medicine, New Haven, Connecticut
  - Nemours / A. I. duPont Hospital for Children, Wilmington, Delaware
  - Golisano Childrens Hospital of Southwest Florida, Fort Myers, Florida
  - Shands Hospital At University Of Florida, Gainesville, Florida
  - Nemours Children'S Clinic, Jacksonville, Florida
  - Nemours Children'S Clinic - Orlando, Orlando, Florida
  - Nemours Children'S Clinic-Pensacola, Pensacola, Florida
  - All Childrens Hospital Specialty Physicians, St. Petersburg, Florida
  - St. Marys Medical Center, West Palm Beach, Florida
  - Childrens Healthcare Of Atlanta - E, Atlanta, Georgia
  - Navicent Health Physician Group, Macon, Georgia
  - St. Luke'S Mountain State Tumor Institute, Boise, Idaho
  - Children'S Center For Cancer And Blood Diseases, Indianapolis, Indiana
  - Blank Childrens Hospital, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - University Of Louisville, Louisville, Kentucky
  - Childrens Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Sinai Hospital Of Baltimore, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - University Of Michigan Cancer Center, Ann Arbor, Michigan
  - Childrens Hospitals And Clinics Of Minnesota, Minneapolis, Minnesota
  - University Of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - University Of Mississippi Medical Center, Jackson, Mississippi
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Valerie Fund Children's Center at St. Joseph's Children's Hospital, Paterson, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - University Of Rochester General Clinical Research Center, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - Unv. Of Nc At Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Akron Children'S Hospital, Akron, Ohio
  - Cincinnati Children'S Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals, Cleveland, Ohio
  - Nationwide Children'S Hospital, Columbus, Ohio
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Childrens Hospital Of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital Of Pittsburgh Of UPMC, Pittsburgh, Pennsylvania
  - Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Monroe Carell Jr Children'S Hosp. At Vanderbilt Tower, Nashville, Tennessee
  - Dell Children'S Medical Center Of Central Texas, Austin, Texas
  - Driscoll Children'S Hospital, Corpus Christi, Texas
  - Texas Children's Cancer and Hematology Centers, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - Scott & White - McLane Children's Specialty Clinic, Temple, Texas
  - Providence Sacred Heart Medical Center, Spokane, Washington
  - MultiCare Institute for Research & Innovation, Tacoma, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Local Institution, New Lambton Heights, New South Wales
  - Queensland Children's Hospital, Sth Brisbane, Queensland
  - Monash Medical Centre Clayton, Clayton, Victoria
  - Local Institution, Parkville, Victoria
- Belgium (4):
  - Local Institution, Brussels
  - Local Institution, Edegem
  - Local Institution, Ghent
  - Local Institution, Leuven
- Canada (5):
  - Alberta Children'S Hospital, Calgary, Alberta
  - Local Institution, Edmonton, Alberta
  - Local Institution, St. John's, Newfoundland and Labrador
  - Children'S Hospital London Health Sciences Centre, London, Ontario
  - Children'S Hospital Of Eastern Ontario, Ottawa, Ontario
- Klinika detske onkologie, Brno, Czechia
- Hungary (3):
  - Local Institution, Budapest
  - Local Institution, Debrecen
  - Local Institution, Pécs
- Mexico (3):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Df, Mexico City
  - Local Institution, Monterrey, Nuevo León
- Local Institution, Christchurch, New Zealand
- Poland (2):
  - Klinika Transplantacji Szpiku Onkologii i Hematologii Dzieciecej, Wroclaw
  - Oddzial Hematologii i Onkologii Dzieciecej, Zabrze
- Local Institution, Caguas, Puerto Rico
- Russia (3):
  - Local Institution, Kirov
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
- Local Institution, Seoul, South Korea

REFERENCES:
- [Derived] Rodriguez V, O'Brien SH, Orgel E, Schultz CL, Esbenshade AJ, Memaj A, Dyme JL, Favatella NA, Mitchell LG. Safety and efficacy of apixaban thrombosis prevention in pediatric patients with obesity and acute lymphoblastic leukemia. Blood Adv. 2025 Sep 23;9(18):4738-4747. doi: 10.1182/bloodadvances.2025016160. PMID 40505060
- [Derived] O'Brien SH, Rodriguez V, Lew G, Newburger JW, Schultz CL, Orgel E, Derr K, Ranalli MA, Esbenshade AJ, Hochberg J, Kang HJ, Dinikina Y, Mills D, Donovan M, Dyme JL, Favatella NA, Mitchell LG; PREVAPIX-ALL investigators. Apixaban versus no anticoagulation for the prevention of venous thromboembolism in children with newly diagnosed acute lymphoblastic leukaemia or lymphoma (PREVAPIX-ALL): a phase 3, open-label, randomised, controlled trial. Lancet Haematol. 2024 Jan;11(1):e27-e37. doi: 10.1016/S2352-3026(23)00314-9. Epub 2023 Nov 16. PMID 37980924
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 512 participants were randomized. 256 is the number of subjects who randomized to each of Apixaban or Standard of Care arm respectively.
Groups:
- Apixaban: Participants will be administered apixaban twice daily by mouth or via a NGT or GT according to weight range during approximately 28 days of induction chemotherapy including asparaginase.
  Weight range - Dose
  >/=35 kg - 2.5 mg twice daily <35 to 25 kg - 2 mg twice daily <25 to 18 kg - 1.5 mg twice daily <18 to 10.5 kg - 1 mg twice daily <10.5 to 6 kg - 0.5 mg twice daily
- Standard of Care: No systemic anticoagulant prophylaxis during induction chemotherapy
Period: Overall Study
Arm/Group | Apixaban | Standard of Care
Started | 256 | 256
Adverse Event Analysis Population | 250 (Out of the 256 participants randomized to Apixaban only 250 participants received an apixaban dose.) | 262 (The 6 subjects who were randomized to apixaban but received no dose were analyzed in Standard of Care.)
Completed | 242 | 249
Not Completed | 14 | 7
Not completed — Lost to Follow-up | 0 | 1
Not completed — Administrative reason by sponsor | 0 | 1
Not completed — Death | 1 | 2
Not completed — Participant withdrew consent | 13 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Apixaban | Standard of Care | Total
Number analyzed (Participants) | 256 | 256 | 512
Age, Continuous [Mean (Standard Deviation); unit: Years] | 7.2 (4.34) | 7.1 (4.39) | 7.2 (4.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 107 | 222
  Male | 141 | 149 | 290
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 59 | 63 | 122
  Not Hispanic or Latino | 196 | 192 | 388
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 25 | 27 | 52
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 12 | 12 | 24
  White | 194 | 194 | 388
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Non-Fatal DVT, PE, and CVST, and VTE-Related-Death
Description: The number of participants with non-fatal deep vein thromboses (DVT) (including asymptomatic and symptomatic), pulmonary embolism (PE), cerebral venous sinus thrombosis (CVST); and venous thromboembolism (VTE) related-death objectively confirmed by a blinded, independent adjudication committee.
  Symptomatic events are included during the intended treatment period. Asymptomatic events are included from scans up to Day 40.
Time Frame: From first dose up to approximately 40 days after first dose
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Standard of Care
Number analyzed (Participants) | 256 | 256
Participants | 31 | 45
Statistical Analysis 1: Comparison: Apixaban vs Standard of Care; Test type: Superiority; p = 0.0403, Cochran-Mantel-Haenszel

2. Primary Outcome: The Number of Participants With Adjudicated Major Bleeding
Description: The number of participants with major bleeding adjudicated by a blinded, independent adjudication committee. Adjudicated major bleeding is defined as bleeding that satisfies one or more of the following criteria:
  1. fatal bleeding
  2. clinically overt bleeding associated with a decrease in hemoglobin of at least 20g/L (ie, 2g/dL) in a 24-hour period
  3. bleeding that is retroperitoneal, pulmonary, intracranial, or otherwise involves the CNS; and/or
  4. bleeding that requires surgical intervention in an operating suite, including interventional radiology.
Time Frame: From first dose up to approximately 34 days after first dose
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Standard of Care
Number analyzed (Participants) | 256 | 256
Participants | 2 | 2
Statistical Analysis 1: Comparison: Apixaban vs Standard of Care; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel

3. Secondary Outcome: The Number of Participants With Non-fatal Asymptomatic Deep Vein Thromboses (DVT)
Description: The number of participants with non-fatal asymptomatic deep vein thromboses (DVT) adjudicated by a blinded, independent adjudication committee
Time Frame: From first dose up to approximately 40 days after first dose
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Standard of Care
Number analyzed (Participants) | 256 | 256
Participants | 27 | 38

4. Secondary Outcome: The Number of Participants With Non-fatal Symptomatic Deep Vein Thromboses (DVT)
Description: The number of participants with non-fatal symptomatic deep vein thromboses (DVT) adjudicated by a blinded, independent adjudication committee
Time Frame: From first dose up to approximately 34 days after first dose
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Standard of Care
Number analyzed (Participants) | 256 | 256
Participants | 4 | 6

5. Secondary Outcome: The Number of Participants With Non-fatal Pulmonary Embolism (PE)
Description: The number of participants with non-fatal pulmonary embolism (PE) adjudicated by a blinded, independent adjudication committee
Time Frame: From first dose up to approximately 34 days after first dose
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Standard of Care
Number analyzed (Participants) | 256 | 256
Participants | 0 | 0

6. Secondary Outcome: The Number of Participants With Cerebral Venous Sinus Thrombosis (CVST)
Description: The number of participants with cerebral venous sinus thrombosis (CVST) adjudicated by a blinded, independent adjudication committee
Time Frame: From first dose up to approximately 34 days after first dose
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Standard of Care
Number analyzed (Participants) | 256 | 256
Participants | 0 | 1

7. Secondary Outcome: The Number of Participants With Venous Thromboembolism (VTE)-Related-death
Description: The number of participants with venous thromboembolism (VTE)-related-death adjudicated by a blinded, independent adjudication committee
Time Frame: From first dose up to approximately 34 days after first dose
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Standard of Care
Number analyzed (Participants) | 256 | 256
Participants | 0 | 0

8. Secondary Outcome: The Number of Participants With Major and Clinically Relevant Non-Major Bleeding (CRNMB)
Description: The number of participants with major and clinically relevant non-major bleeding (CRNMB) adjudicated by a blinded, independent adjudication committee
  CRNM bleeding is defined as bleeding that satisfies one or both of the following:
  1. overt bleeding for which blood product is administered and not directly attributable to the subject's underlying medical condition and
  2. bleeding that requires medical or surgical intervention to restore hemostasis, other than in an operating room
Time Frame: From first dose up to approximately 34 days after first dose
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Standard of Care
Number analyzed (Participants) | 256 | 256
Participants | 13 | 5

9. Secondary Outcome: The Number of Participant Deaths
Description: The number of participant deaths adjudicated by a blinded, independent adjudication committee
Time Frame: From first dose date until the end of the treatment period + 30 days (Up to approximately 59 days)
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Standard of Care
Number analyzed (Participants) | 256 | 256
Participants | 1 | 3

10. Secondary Outcome: The Number of Participants With an Arterial Thromboembolic Event
Description: The number of participants with an arterial thromboembolic event including paradoxical embolism and stroke adjudicated by a blinded, independent adjudication committee
Time Frame: From first dose up to approximately 34 days after first dose
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Standard of Care
Number analyzed (Participants) | 256 | 256
Participants | 0 | 0

11. Secondary Outcome: The Number of Participants With a CVAD-Related Infection
Description: The number of participants with a central venous access device (CVAD)-related infection adjudicated by a blinded, independent adjudication committee
Time Frame: From first dose up to approximately 34 days after first dose
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Standard of Care
Number analyzed (Participants) | 256 | 256
Participants | 1 | 6

12. Secondary Outcome: The Number of Participants Needing Catheter Replacements During the Study
Description: The number of participants needing catheter replacements during the study
Time Frame: From first dose up to approximately 34 days after first dose
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Standard of Care
Number analyzed (Participants) | 256 | 256
Participants | 3 | 2

13. Secondary Outcome: The Number of Participants With CVAD Patency Restoration Events After Thrombolytic Therapy Use
Description: The number of participants with central venous access device (CVAD) patency restoration events after thrombolytic therapy use
Time Frame: From first dose up to approximately 34 days after first dose
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Standard of Care
Number analyzed (Participants) | 256 | 256
Participants | 0 | 0

14. Secondary Outcome: The Number Participants Experiencing Superficial Vein Thrombosis Events
Description: The number participants experiencing superficial vein thrombosis events.
  Clots that occur in a superficial vein ie, cephalic vein, basilic vein (upper extremity) or saphenous vein (lower extremity) confirmed by radiographic imaging.
Time Frame: From first dose up to approximately 34 days after first dose
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Standard of Care
Number analyzed (Participants) | 256 | 256
Participants | 4 | 2

15. Secondary Outcome: The Number of Participants With Clinically Relevant Non-Major Bleeding Events (CRNMB)
Description: The number of participants with clinically relevant non-major bleeding events (CRNMB) adjudicated by a blinded, independent adjudication committee.
  CRNM bleeding is defined as bleeding that satisfies one or both of the following:
  1. overt bleeding for which blood product is administered and not directly attributable to the subject's underlying medical condition and
  2. bleeding that requires medical or surgical intervention to restore hemostasis, other than in an operating room
Time Frame: From first dose up to approximately 34 days after first dose
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Standard of Care
Number analyzed (Participants) | 256 | 256
Participants | 11 | 3

16. Secondary Outcome: The Number of Participants With Minor Bleeding Events
Description: The number of participants with minor bleeding events adjudicated by a blinded, independent adjudication committee.
  Minor bleeding defined as any overt or macroscopic evidence of bleeding that does not fulfill the criteria for either major bleeding or CRNMB
Time Frame: From first dose up to approximately 34 days after first dose
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Standard of Care
Number analyzed (Participants) | 256 | 256
Participants | 37 | 20

17. Secondary Outcome: The Number of Platelet Transfusions Needed During the Study
Description: The number of platelet transfusions needed during the study.
  The events are not adjudicated. A subject could have more than one platelet transfusion.
Time Frame: From first dose up to approximately 34 days after first dose
Population: All randomized participants
Measure: Number; unit: Platelet Transfusions
Arm/Group | Apixaban | Standard of Care
Number analyzed (Participants) | 256 | 256
Platelet Transfusions | 266 | 248

18. Secondary Outcome: Maximum Observed Concentration (Cmax)
Description: The maximum observed concentration (Cmax) was measured to assess the pharmacokinetics of oral or enteric apixaban in pediatric subjects receiving induction chemotherapy.
Time Frame: pre-dose, 1-4 hours post dose
Population: All randomized participants in the apixaban arm with available pharmacokinetic data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Participants Weight Range ≥ 35 kg: Participants will be administered 2.5mg apixaban twice daily by mouth or via a NGT or GT according to weight range during approximately 28 days of induction chemotherapy including asparaginase
- Participants Weight Range 25 to < 35 kg: Participants will be administered 2mg apixaban twice daily by mouth or via a NGT or GT according to weight range during approximately 28 days of induction chemotherapy including asparaginase
- Participants Weight Range 18 to < 25 kg: Participants will be administered 1.5mg apixaban twice daily by mouth or via a NGT or GT according to weight range during approximately 28 days of induction chemotherapy including asparaginase
- Participants Weight Range 10.5 to < 18 kg: Participants will be administered 1mg apixaban twice daily by mouth or via a NGT or GT according to weight range during approximately 28 days of induction chemotherapy including asparaginase
Arm/Group | Participants Weight Range ≥ 35 kg | Participants Weight Range 25 to < 35 kg | Participants Weight Range 18 to < 25 kg | Participants Weight Range 10.5 to < 18 kg
Number analyzed (Participants) | 71 | 30 | 50 | 73
ng/mL | 56.5 (36.5) | 63.6 (38.6) | 61.4 (43.9) | 54.2 (46.8)

19. Secondary Outcome: Trough Observed Concentration (Cmin)
Description: The trough observed concentration (Cmin) was measured to assess the pharmacokinetics of oral or enteric apixaban in pediatric subjects receiving induction chemotherapy.
Time Frame: pre-dose, 1-4 hours post dose
Population: All randomized participants in the apixaban arm with available pharmacokinetic data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Participants Weight Range ≥ 35 kg | Participants Weight Range 25 to < 35 kg | Participants Weight Range 18 to < 25 kg | Participants Weight Range 10.5 to < 18 kg
Number analyzed (Participants) | 71 | 30 | 50 | 73
ng/mL | 18.8 (57.8) | 18.1 (97.4) | 12 (142) | 12.9 (113)

20. Secondary Outcome: Area Under the Concentration-Time Curve [AUC(TAU)]
Description: The area under the concentration-time curve [AUC(TAU)] was measured to assess the pharmacokinetics of oral or enteric apixaban in pediatric subjects receiving induction chemotherapy.
Time Frame: pre-dose, 1-4 hours post dose
Population: All randomized participants in the apixaban arm with available pharmacokinetic data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•h/mL
Arm/Group | Participants Weight Range ≥ 35 kg | Participants Weight Range 25 to < 35 kg | Participants Weight Range 18 to < 25 kg | Participants Weight Range 10.5 to < 18 kg
Number analyzed (Participants) | 71 | 30 | 50 | 73
ng•h/mL | 470 (35.3) | 510 (42.7) | 453 (44.8) | 416 (48.5)

21. Secondary Outcome: Anti-FXa Activity
Description: Anti-FXa Activity was measured to characterize the relationship between apixaban plasma concentration and anti-FXa activity in pediatric subjects receiving induction chemotherapy
Time Frame: pre-dose and 2.5 hours after dosing on day 7. Day 8 and day 15.
Population: All randomized participants in the apixaban arm with available pharmacodynamic data
Measure: Mean (Standard Deviation); unit: Anti-FXa activity (ng/mL)
Arm/Group | Participants Weight Range ≥ 35 kg | Participants Weight Range 25 to < 35 kg | Participants Weight Range 18 to < 25 kg | Participants Weight Range 10.5 to < 18 kg
Number analyzed (Participants) | 28 | 14 | 21 | 31
Anti-FXa activity (ng/mL)
  Day 7 (Predose): number analyzed (Participants) | 9 | 5 | 6 | 12
  Day 7 (Predose) | 55.3 (16.4) | 62.2 (19.4) | 52.8 (16) | 44.2 (12.9)
  Day 7 (2.5 hours): number analyzed (Participants) | 23 | 14 | 21 | 31
  Day 7 (2.5 hours) | 78.7 (28.8) | 72.1 (30.6) | 77.5 (30.8) | 87.5 (45.5)
  Day 8: number analyzed (Participants) | 4 | 0 | 2 | 2
  Day 8 | 55.2 (8.96) |  | 47.5 (10.6) | 48 (11.3)
  Day 15: number analyzed (Participants) | 28 | 10 | 17 | 26
  Day 15 | 70.2 (28) | 75.3 (33.9) | 63.9 (21.6) | 64.8 (25.3)

ADVERSE EVENTS:
Time Frame: AEs are collected from the first dose date until the end of the treatment period + 2 days (Up to approximately 31 days) SAEs are collected from the first dose date until the end of the treatment period + 30 days (Up to approximately 59 days). All Cause Mortality was collected from first dose up to DBL date: Sep-13-2021 (up to approximately 6 years.)
Groups:
- Apixaban: Participants will be administered apixaban twice daily by mouth or via a NGT or GT according to weight range during approximately 28 days of induction chemotherapy including asparaginase
Arm/Group | Apixaban | Standard of Care
All-Cause Mortality (participants affected / at risk) | 1/250 | 4/262
Serious Adverse Events (participants affected / at risk) | 91/250 | 83/262
Other Adverse Events (participants affected / at risk) | 204/250 | 193/262
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban (N=250) | Standard of Care (N=262)
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Coagulopathy (Blood and lymphatic system disorders) | 1 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 15 | 16
Neutropenia (Blood and lymphatic system disorders) | 0 | 3
Cardiac arrest (Cardiac disorders) | 1 | 1
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Pneumopericardium (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Ocular hypertension (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Colitis (Gastrointestinal disorders) | 2 | 5
Constipation (Gastrointestinal disorders) | 1 | 5
Haematochezia (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 3
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 3
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Device related thrombosis (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 7 | 7
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 2
Hypersensitivity (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 2
Aspergillus infection (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 3 | 2
Enterocolitis infectious (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 1 | 0
Fungal sepsis (Infections and infestations) | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 1
Haemophilus bacteraemia (Infections and infestations) | 1 | 0
Infective thrombosis (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 2 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 3
Postoperative wound infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 6 | 5
Septic shock (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Stomatococcal infection (Infections and infestations) | 0 | 1
Streptococcal sepsis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Epidural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Meningitis chemical (Injury, poisoning and procedural complications) | 1 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Human rhinovirus test positive (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 4
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebral venous sinus thrombosis (Nervous system disorders) | 0 | 3
Encephalopathy (Nervous system disorders) | 0 | 2
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Leukoencephalopathy (Nervous system disorders) | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 2
Seizure (Nervous system disorders) | 2 | 2
Syncope (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 1
Testicular cyst (Reproductive system and breast disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 6
Embolism (Vascular disorders) | 9 | 3
Hypertension (Vascular disorders) | 3 | 0
Hypotension (Vascular disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 2
Subclavian vein thrombosis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 2 | 1
Venous thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban (N=250) | Standard of Care (N=262)
Anaemia (Blood and lymphatic system disorders) | 85 | 88
Febrile neutropenia (Blood and lymphatic system disorders) | 14 | 7
Neutropenia (Blood and lymphatic system disorders) | 17 | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 28 | 25
Tachycardia (Cardiac disorders) | 15 | 13
Abdominal distension (Gastrointestinal disorders) | 17 | 12
Abdominal pain (Gastrointestinal disorders) | 34 | 48
Constipation (Gastrointestinal disorders) | 58 | 50
Diarrhoea (Gastrointestinal disorders) | 26 | 16
Nausea (Gastrointestinal disorders) | 16 | 20
Stomatitis (Gastrointestinal disorders) | 12 | 15
Vomiting (Gastrointestinal disorders) | 18 | 17
Fatigue (General disorders) | 14 | 20
Pyrexia (General disorders) | 13 | 11
Alanine aminotransferase increased (Investigations) | 46 | 39
Aspartate aminotransferase increased (Investigations) | 28 | 18
Blood bilirubin increased (Investigations) | 17 | 16
Neutrophil count decreased (Investigations) | 22 | 26
Platelet count decreased (Investigations) | 54 | 55
White blood cell count decreased (Investigations) | 21 | 28
Hyperglycaemia (Metabolism and nutrition disorders) | 19 | 30
Hypoalbuminaemia (Metabolism and nutrition disorders) | 29 | 34
Hypocalcaemia (Metabolism and nutrition disorders) | 12 | 21
Hyponatraemia (Metabolism and nutrition disorders) | 36 | 30
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 19
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28 | 25
Pain in jaw (Musculoskeletal and connective tissue disorders) | 14 | 15
Headache (Nervous system disorders) | 16 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 24 | 14
Hypertension (Vascular disorders) | 23 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/53/NCT02369653/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/53/NCT02369653/SAP_001.pdf